CLINICAL TRIAL: NCT02325102
Title: Potential Clinical and Biological Effects of Viral and Bacterial Co-infections in Otherwise Healthy Children in Pediatric Department
Brief Title: Effects of Viral and Bacterial Co-infections in Otherwise Healthy Children Hospitalized in Pediatric Department
Status: Completed | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HMC102-13
Record Dates: First submitted 2014-12-02; First posted 2014-12-24 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Coinfection
MeSH Terms: conditions — Coinfection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention — As this is an observational study, no intervention was conducted.

SUMMARY:
Co-occurence of multiple pathogens in children is a known phenomenon, however the potential effect on the probability to develop a disease and on its severity, as well as the relationships between them, has not been studied adequately.

In this study, children admitted to the pediatric department with a clinical presentation of an infectious disease were tested for the presence of multiple pathogens. Data about their clinical status and about the accessory examinations performed during hospitalization were collected and analyzed.

DETAILED DESCRIPTION:
Introduction The relationship between viral and bacterial infections in the respiratory tract in children has long been learnt and documented in the medical literature. A large scale American study which was held during the "swine flu" (influenza A H1N1) pandemic in 2009-2010 documented pneumonia (or other pulmonary infection) of bacterial source in one third of the patients admitted to intensive care units (PICU - Pediatric Intensive Care Unit) [1]. Similar data and even higher incidence rates also exist for bronchiolitis caused by RSV (respiratory syncytial virus) [2]. These and similar studies raise questions about the real need for antibiotic treatment and whether it is being judiciously prescribed (as it turned out, for example, that there are places in the world where 30-90% of the viral bronchiolitis cases are treated with antibiotics [3]), which puts the patient at risk for side effects and potentially increases bacterial resistance. Moreover, one cannot ignore the fact that otherwise healthy children and children with comorbidity (such as chronic carrier state or relevant background disease) are not always being addressed separately in these studies. Despite all this, there is consensus that children with respiratory viral disease, mainly one that requires hospitalization in PICU, will benefit from empirical antibiotic treatment [4, 5]. On the other hand, when it comes to the potential impact of antiviral treatment on the course of a pulmonary bacterial disease during infection with influenza virus, the results are not encouraging, but the seasonal vaccination plays a key role in reducing the above morbidity [6]. As to whether the presence of a viral infection at the same time affects the severity of pulmonary bacterial infection (i.e. The disease is more serious than that of a viral origin only), there is evidence demonstrating an increase in mortality, duration of mechanical ventilation and duration of hospitalization in mixed bacterial and viral disease [7]. Several studies found and isolated some viruses of different types in the same respiratory ailment, but unanimity as to whether there is correlation between the number of viruses and the severity of the disease is missing [8, 9].

In addition to the multiplicity of sources dealing with the link between viral and bacterial respiratory infections, especially influenza and RSV, there is recent evidence in the literature of a viral-bacterial etiology in acute otitis media [10, 11], but so far a limited number of works has been made about the same relationship of other viruses or in other systems.

The goals of this article:

1. To determine whether the data available in the context of mixed infections in respiratory diseases (see above) are also valid for diseases in other body systems.
2. To discover whether the relationship between viral and bacterial infection is as strong as in the respiratory system
3. to study the impact of the co-infection on morbidity (severity, length of stay, complications)
4. to link between specific infection and its common mixed pathogens
5. to specify age sections, gender, demographic characteristics, clinical condition, at which co-infections (and relevant consequences) predominate

Methods The study group comprised currently or recently febrile, otherwise healthy children aged 0 to 17 years admitted at several medical centers (Hillel Yaffe, Bnai Zion) in Israel, who were found to have viral, bacterial or both infections. Exclusion criteria are listed below (Table 1).

When a child meeting the above criteria was admitted, parent (or child's legal custodian) were given verbal and written explanation by a clinical investigator, signed an informed consent and approved him to collect blood samples and nasal or rectal swab. In accordance to the clinical presentation, additional tests were performed and included blood, urine and stool cultures and some viral and bacterial serologies.

For each patient, individual history was taken; presenting symptoms, physical examinations and lab results were documented; and additional data such as antibiotic therapy, length of stay and complications were collected during hospitalization by authorized medical staff using standard techniques and methods.

Specimen sampling:

* Nasal swab
* Blood sampling with CBC and chemistry tubes
* Rectal swab (only in case of diarrhea)

Laboratory procedures:

Specimens were immediately placed in a refrigerator at 4°C, transferred to MeMed laboratory no longer than 5 hours following sampling.

In the laboratory, blood tests included CBC, bacterial and viral PCR incl. ELISA.

Although clinical signs were usually documented in a great detail, this method is problematic and prone bias for the purpose of defining infection, owing to the investigator's individual interpretation. Thus, in this study only microbiological definitions were used. Viral infection was defined as PCR positive for viral genome or as the presence of IgM antibody against viral specific antigen.

Bacterial infection required PCR positive for bacterial genome sequence, or colony counts 105 cfu/ml of diagnostic sample for each single species obtained, or the presence of IgM antibody against bacterial specific.

Data analysis:

All of the above information was transferred to and arranged in a designated database developed and maintained by the sub-investigators.

In the database, the investigators applied the exclusion criteria, found all patients with viral and bacterial co-infections and analyzed the investigated variants.

Table 1: Exclusion Criteria Afebrile for more than 72 hours

Chronic illness Immune compromised (due to immunosuppressive drugs, neoplastic disease, etc.) History of prematurity or IUGR Not fully vaccinated for age according to national routine vaccination program

Infection not being the primary diagnosis

Under antibiotic therapy:

Currently receiving Recently received (less than 48 hours) No infection was documented during research period

ELIGIBILITY:
Inclusion Criteria:

* Currently or recently febrile, otherwise healthy children aged 0 to 17 years admitted at several medical centers (Hillel Yaffe, Bnai Zion) in Israel, who were found to have viral, bacterial or both infections.

Exclusion Criteria:

* Afebrile for more than 72 hours
* Chronic illness
* Immune compromised (due to immunosuppressive drugs, neoplastic disease, etc.)
* History of prematurity or IUGR
* Not fully vaccinated for age according to national routine vaccination program
* Infection not being the primary diagnosis
* Under antibiotic therapy:
* Currently receiving
* Recently received (less than 48 hours)
* No infection was documented during research period

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: otherwise healthy children admitted in pediatric department
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
number of patients with co-infections | 2 years
  Patients in whom 2 or more pathogens were found in culture, serology or other tests.

SECONDARY OUTCOMES:
Types and species of pathogens | 2 years

OTHER OUTCOMES:
Inflammation indicators in lab results of each patient | 2 years
  WBC count and differential, CRP, ESR

CONTACTS AND LOCATIONS:
Overall Officials: Nitai A Levy, MD, Principal Investigator — Physician

REFERENCES:
- [Background] Randolph AG, Vaughn F, Sullivan R, Rubinson L, Thompson BT, Yoon G, Smoot E, Rice TW, Loftis LL, Helfaer M, Doctor A, Paden M, Flori H, Babbitt C, Graciano AL, Gedeit R, Sanders RC, Giuliano JS, Zimmerman J, Uyeki TM; Pediatric Acute Lung Injury and Sepsis Investigator's Network and the National Heart, Lung, and Blood Institute ARDS Clinical Trials Network. Critically ill children during the 2009-2010 influenza pandemic in the United States. Pediatrics. 2011 Dec;128(6):e1450-8. doi: 10.1542/peds.2011-0774. Epub 2011 Nov 7. PMID 22065262
- [Background] Thorburn K, Harigopal S, Reddy V, Taylor N, van Saene HK. High incidence of pulmonary bacterial co-infection in children with severe respiratory syncytial virus (RSV) bronchiolitis. Thorax. 2006 Jul;61(7):611-5. doi: 10.1136/thx.2005.048397. Epub 2006 Mar 14. PMID 16537670
- [Background] Spurling GK, Fonseka K, Doust J, Del Mar C. Antibiotics for bronchiolitis in children. Cochrane Database Syst Rev. 2007 Jan 24;(1):CD005189. doi: 10.1002/14651858.CD005189.pub2. PMID 17253545
- [Background] Levin D, Tribuzio M, Green-Wrzesinki T, Ames B, Radwan S, Jarvis JD, Vaccaro T, Modlin JF. Empiric antibiotics are justified for infants with respiratory syncytial virus lower respiratory tract infection presenting with respiratory failure: a prospective study and evidence review. Pediatr Crit Care Med. 2010 May;11(3):390-5. doi: 10.1097/PCC.0b013e3181b809c5. PMID 19838143
- [Background] American Academy of Pediatrics Subcommittee on Diagnosis and Management of Bronchiolitis. Diagnosis and management of bronchiolitis. Pediatrics. 2006 Oct;118(4):1774-93. doi: 10.1542/peds.2006-2223. PMID 17015575